CLINICAL TRIAL: NCT04486612
Title: Department of Anesthesiology and Reanimation, Faculty of Medicine, Osmangazi University, Eskişehir, Turkey
Brief Title: Ultrasonographic Measurement of Internal Jugular Vein as a Predictor of Hypotension Following Spinal Anesthesia
Acronym: IJV
Status: Completed | Type: Observational
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Yeliz KILIÇ, Assistant Professor, Eskisehir Osmangazi University
Other Study IDs: 10.12.19/43
Record Dates: First submitted 2020-07-22; First posted 2020-07-24 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Spinal Anesthetics Causing Adverse Effects in Therapeutic Use; Hypotension Postprocedural
Keywords: spinal anesthesia; internal jugular vein; hypotension; ultrasonography
MeSH Terms: conditions — Hypotension | interventions — Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hypotension
  Interventions: Other: spinal anesthesia
- non-hypotension
  Interventions: Other: spinal anesthesia

INTERVENTIONS:
Other: spinal anesthesia — prospective observational study

SUMMARY:
Hypotension after spinal anesthesia is associated with significant perioperative morbidity and mortality, especially in hypovolemic patients. Ultrasonographic measurement of internal jugular vein (IJV) has been recently shown as effective in predicting the intravascular volume status. The aim was to investigate the reliability of preanesthetic ultrasound measurements of IJV in predicting hypotension after spinal anesthesia.

DETAILED DESCRIPTION:
Hypotension after spinal anesthesia is associated with significant perioperative morbidity and mortality, especially in hypovolemic patients. Ultrasonographic measurement of internal jugular vein (IJV) has been recently shown as effective in predicting the intravascular volume status. The aim was to investigate the reliability of preanesthetic ultrasound measurements of IJV in predicting hypotension after spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-65 Patients who read and accept the consent form of the study Patients undergoing elective surgery under spinal anesthesia

Exclusion Criteria:

* under 18 years old, ASA scores 3-4, presence of any significant hepatic, renal, cardiavasculary, or respiratory disease, having left ventricular ejection fraction less than 40%, and allergy to study medications.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18-65
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-24 (Actual)

PRIMARY OUTCOMES:
The association between sonographic measurements and postspinal hypotension | first 30 minute
  The aim of the study is to evaluate the association between sonographic measurements and postinduction hypotension.

CONTACTS AND LOCATIONS:
Overall Officials: yeliz kılıç, Ass. Prof, Principal Investigator — Eskişehir Osmangazi Univercity
Locations (1):
- Eskişehir Osmangazi Univercity, Eskişehir, Turkey (Türkiye)